CLINICAL TRIAL: NCT04541498
Title: Impact of Air Pollution and Climate Changes on the Epidemiology of Cardiovascular Disease
Acronym: PL-PARTICLES
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lukasz Kuzma, MD, PhD, Medical University of Bialystok
Other Study IDs: UMB-KKI-103
Record Dates: First submitted 2020-08-21; First posted 2020-09-09 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-09

CONDITIONS: Pollution; Exposure; Acute Coronary Syndrome; Chronic Coronary Insufficiency; Particulate Matter Inhalation Injury; Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Air pollution; Particulate Matter; Acute Coronary Syndromes; Cardiovascular Disease; Risk factors
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases | interventions — Climate Change

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population of Poland: Exposure to short term long term effects of air pollution and climate change
  Interventions: Other: Impact of air pollution and climate changes
- Patients with Acute Coronary and Cerebral Syndromes: Exposure to short term long term effects of air pollution and climate change
  Interventions: Other: Impact of air pollution and climate changes

INTERVENTIONS:
Other: Impact of air pollution and climate changes — To assess the short- and long- term impact of air pollution and climate changes

SUMMARY:
Despite the fact that the topic of air pollution has been in focus of researchers for many years, there are no big studies that take up the matter of its influence on acute coronary, cerebral syndromes and CVD mortality in Europe. Taking into consideration the scarce number of surveys from Europe the investigators decided to analyze the impact of air pollution on cardiovascular diseases and CVD mortality in Poland.

DETAILED DESCRIPTION:
Air quality and its impact on health was put in the spotlight since the infamous Great Smog of London. Since then, it became clear that adverse effects are serious and can no longer be ignored. According to the World Health Organization (WHO) estimations, in last year ambient air pollution caused 4,200,000 deaths worldwide. These statistics included a total of 29,165 deaths that were attributed to air pollution in Poland.

The vast of studies are conducted in highly polluted areas, in which patients are exposed to extreme concentrations like China oraz Indie. Taking into consideration the scarce number of surveys from Europe the investigators decided to analyze the impact of air pollution and cardiovascular diseases in Poland.

Data on morbidity and mortality were collected from the National Statistical Office in Poland. The data of air pollutions and gases were obtained from Voivodeship Inspectorate for Environmental Protection. The daily meteorological data were obtained from the Institute of Meteorology and Water Manageme

ELIGIBILITY:
Inclusion criteria:

- residents from analysed area.

Exclusion criteria

- none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In primary we focus on Podlaskie Voivodeship. The region is located in north-east Poland which is a developing country as well as one of the poorest regions of the EU. Within four national parks, the region is widely known as the Green Lungs of Poland, mainly due to large areas covered by forests, lack of factories, and relatively low industrialization.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of acute coronary syndromes | Through study completion, an average of 1 year
  Number of acute coronary syndromes related with impact of air pollution
Incidence of cardiovascular mortality | Through study completion, an average of 1 year
  Number of cardiovascular deaths related with impact of air pollution
Incidence of acute cerebral syndromes | Through study completion, an average of 1 year
  Number of acute cerebral syndromes related with impact of air pollution

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Kuzma, MD, PhD, Principal Investigator — Medical University of Bialystok, Department of Invasive Cardiology
Locations (1):
- Department of Invasive Cardiology Medical University of Białystok 24A M. Skłodowskiej-Curie St., Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication

REFERENCES:
- [Result] Kuzma L, Pogorzelski S, Struniawski K, Dobrzycki S, Bachorzewska-Gajewska H. Effect of air pollution on the number of hospital admissions for acute coronary syndrome in elderly patients. Pol Arch Intern Med. 2020 Jan 31;130(1):38-46. doi: 10.20452/pamw.15064. Epub 2019 Nov 19. PMID 31742576
- [Result] Kuzma L, Pogorzelski S, Struniawski K, Bachorzewska-Gajewska H, Dobrzycki S. Exposure to air pollution-a trigger for myocardial infarction? A nine-year study in Bialystok-the capital of the Green Lungs of Poland (BIA-ACS registry). Int J Hyg Environ Health. 2020 Aug;229:113578. doi: 10.1016/j.ijheh.2020.113578. Epub 2020 Aug 3. PMID 32758862
- [Result] Kuzma L, Struniawski K, Pogorzelski S, Bachorzewska-Gajewska H, Dobrzycki S. Gender Differences in Association between Air Pollution and Daily Mortality in the Capital of the Green Lungs of Poland-Population-Based Study with 2,953,000 Person-Years of Follow-Up. J Clin Med. 2020 Jul 23;9(8):2351. doi: 10.3390/jcm9082351. PMID 32717977
- [Result] Kuzma L, Wanha W, Kralisz P, Kazmierski M, Bachorzewska-Gajewska H, Wojakowski W, Dobrzycki S. Impact of short-term air pollution exposure on acute coronary syndrome in two cohorts of industrial and non-industrial areas: A time series regression with 6,000,000 person-years of follow-up (ACS - Air Pollution Study). Environ Res. 2021 Jun;197:111154. doi: 10.1016/j.envres.2021.111154. Epub 2021 Apr 17. PMID 33872649
- [Derived] Rogalska E, Kurasz A, Kuzma L, Bachorzewska-Gajewska H, Dobrzycki S, Kozinski M, Sobkowicz B, Tomaszuk-Kazberuk A. Comparing Atrial-Fibrillation Validated Rapid Scoring Systems in the Long-Term Mortality Prediction in Patients Referred for Elective Coronary Angiography: A Subanalysis of the Bialystok Coronary Project. Int J Environ Res Public Health. 2022 Aug 21;19(16):10419. doi: 10.3390/ijerph191610419. PMID 36012052